# **COVER PAGE**

OFFICIAL TITLE

Effect of Skin-to-Skin Contact on Father-Infant Bonding: A Randomized Controlled Tr

NCT NUMBER

[if available]

DOCUMENT TYPE

Informed Consent Form (ICF) - Adult Fathers

DOCUMENT DATE

18 Jan 2023

UNIQUE PROTOCOL ID

2023-YÖNP-0008

## Informed Consent Form (English Translation)

## INFORMED CONSENT FORM (ENGLISH TRANSLATION)

Study Title: Effect of Skin-to-Skin Contact on Father-Infant Bonding: A Randomized

Controlled Trial

Protocol ID: 2023-YÖNP-0008

Sponsor/Institution: Çanakkale Onsekiz Mart University (ÇOMÜ)

#### Introduction

You are invited to take part in a research study about father-infant skin-to-skin contact. Please read this information carefully. You may ask questions before deciding whether to participate.

## Purpose

To evaluate whether skin-to-skin contact improves bonding between fathers and their newborns.

#### **Procedures**

If you agree, you will be randomly assigned to one of three groups: early one-time skin-to-skin, frequent skin-to-skin, or standard care. You will complete a brief questionnaire at baseline and a follow-up questionnaire at about 3 months postpartum, including the Paternal-Infant Attachment Scale (PIAS). Skin-to-skin involves holding your baby against your bare chest for approximately 15 minutes per session.

#### Risks/Discomforts

Minimal risks are anticipated (e.g., temporary discomfort from holding position). No medical treatment is provided as part of the study.

#### **Benefits**

You may or may not benefit directly. Your participation may help improve understanding of father-infant bonding.

## Confidentiality

Your information will be kept confidential. Study data will be de-identified. Results may be published without identifying you.

#### Voluntary Participation and Withdrawal

Your participation is voluntary. You may withdraw at any time without penalty or loss of benefits to which you are otherwise entitled.

#### Compensation/Costs

There is no payment for participation and no additional costs to you.

## Contacts

If you have questions about the study, please contact the research team. For questions about your rights, you may contact the institutional ethics committee.

## Consent

By signing below, you indicate that you have read and understood this form and agree to participate.

(Signature and date lines to be added on the local consent form.)